CLINICAL TRIAL: NCT02235363
Title: Thread Lift by Use of Retaining Ligaments With V-lock Barbed Sutures : Under the Condition of Using the Tensiometer and FACE-Q
Brief Title: Thread Lift by Use of Retaining Ligaments
Acronym: TL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winners Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thread Lift
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Face Lift; Suspension Technique; Minimal Invasive Surgery
Keywords: face lift; thread lift; retaining ligament; V-Loc sutures; tensiometer; FACE-Q

STUDY DESIGN:
Intervention Model Description: 369 consecutive patients underwent the suture suspension technique, so called thread lift, using 3-0 V-Loc 180 device for facial rejuvenation with (n=305) or without additional facial procedures (n=64). The follow-up period ranged from 22 months to 43 months postoperatively, with a mean of 34.3 months.
Oversight: Data Monitoring Committee: No

ARMS (1):
- facelift (Experimental): In facial rejuvenating surgery, the current trend calls for fewer and less noticeable scars with desired results. Especially to improve the jowls and nasolabial folds, the thread lift is a simple and inexpensive technique for patients who do not wish to undergo the typical facelift surgery, but the weak points of it are less effective and shorter duration than the conventional facelift.The investigators propose the new method of the thread lifting the subdermal and subcutaneous layer by use of the retaining ligaments with two fixation points on both temporal fascia and retaining ligaments.
  Interventions: Procedure: thread lift

INTERVENTIONS:
Procedure: thread lift — In facial rejuvenating surgery, the current trend calls for fewer and less noticeable scars with desired results. Especially to improve the jowls and nasolabial folds, the thread lift is a simple and inexpensive technique for patients who do not wish to undergo the typical facelift surgery, but the weak points of it are less effective and shorter duration than the conventional facelift.The investigators propose the new method of the thread lifting the subdermal and subcutaneous layer by use of the retaining ligaments with two fixation points on both temporal fascia and retaining ligaments.
  Other Names: suspension technique with V-Loc barbed sutures

SUMMARY:
In facial rejuvenating surgery, the current trend calls for fewer and less noticeable scars with desired results. Especially to improve the jowls and nasolabial folds, the thread lift is a simple and inexpensive technique for patients who do not wish to undergo the typical facelift surgery, but the weak points of it are less effective and shorter duration than the conventional facelift.The investigators propose the new method of the thread lifting the subdermal and subcutaneous layer with a fiberoptic needle by use of the retaining ligaments with two fixation points on both temporal fascia and retaining ligaments. For the intraoperative evaluation the tensiometer was applied and for the postoperative evaluation the FACE-Q applied.

DETAILED DESCRIPTION:
In facial rejuvenating surgery, the current trend calls for fewer and less noticeable scars with desired results. Especially to improve the jowls and nasolabial folds, the thread lift is a simple and inexpensive technique for patients who do not wish to undergo the typical facelift surgery, but the weak points of it are less effective and shorter duration than the conventional facelift.The investigators propose the new method of the thread lifting the subdermal and subcutaneous layer with a fiberoptic needle by use of the retaining ligaments.

Retrospective analysis was performed on 369 consecutive patients undergoing the suture suspension technique between January of 2012 and December of 2015, so called thread lift, using 3-0 V-Loc 180 device for facial rejuvenation with (n=305) or without additional facial procedures (n=64). The follow-up period ranged from 22 months to 43 months postoperatively, with a mean of 34.3 months. There are asymmetry(n=2), scar revision(n=1), revision(n=4), dimpling(n=1), suboptimal outcomes(n=9), and stitch abscess(n=1). The thread lift by use of the retaining ligaments with V-lock barbed sutures can be recommended as an alternative technique in the facelift.

ELIGIBILITY:
Inclusion Criteria:

* primary case
* secondary case

Exclusion Criteria:

* wide scar tissue on face
* allergy to foreign body(thread)
* no skin excess

Ages: 23 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Revision or reoperation | 3 and 6 months
  Checking whether revision was done by patients' need or not.

SECONDARY OUTCOMES:
Suboptimal outcomes | 3 and 6 months
  Checking whether patients were satisfied with the postoperative outcomes of their faces or not.
Asymmetry | 3 and 6 months
  Comparing the degree of sagging of the right and left faces to see if there is any difference.
Scar revision | 3 and 6 months
  Checking whether scar revision was done due to hypertrophic scar on the operative sites or not.
Dimpling | 3 and 6 months
  Checking whether patients complained about dimpling on the operation sites of their faces or not.
Stitch abscess | 3 and 6 months
  Checking whether the operative sites were infected or not.

CONTACTS AND LOCATIONS:
Overall Officials: CHEOLHWAN KIM, M.D., Principal Investigator — Winners Clinic
Locations (1):
- The Department of Plastic Surgery, Winners Clinic, Seoul, South Korea

REFERENCES:
- [Background] Sasaki GH, Cohen AT. Meloplication of the malar fat pads by percutaneous cable-suture technique for midface rejuvenation: outcome study (392 cases, 6 years' experience). Plast Reconstr Surg. 2002 Aug;110(2):635-54; discussion 655-7. doi: 10.1097/00006534-200208000-00042. PMID 12142689